CLINICAL TRIAL: NCT04879446
Title: Evaluation Of The Effects Of Advanced Platelet Rich Fibrin And Concenrated Growth Factor Liquids On Dental Implant Osseointegration: A Randomized Controlled Double-Blind Clinical Trial
Brief Title: The Effect of Growth Factor on Implant Osseointegration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uğur Can ÜNLÜGENÇ (Other)
Collaborators: Mustafa Kemal University (Other)
Responsible Party: Sponsor-Investigator, Uğur Can ÜNLÜGENÇ, Researcher, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19.U.019
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Bone Loss, Alveolar; Resorption, Bone; Osseointegration Failure of Dental Implant
Keywords: Advanced Platelet Rich Fibrin; Concentrated Growth Factor; Implant Osseointegration; Resonance Frequency Analysis
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption

STUDY DESIGN:
Intervention Model Description: This is a split-mouth design study. This study evaluating the effects of advanced platelet-rich fibrin and concentrated growth factor liquids on dental implant osseointegration was planned as a randomized, clinical controlled and prospective study. A total of 32 patients included in our study were divided into two groups of 16. It was planned to apply 2 implants to each patient and to evaluate each patient as one side as the control and the other as the study group. In other words, while there was a study group and a control group in the CGF group, there was also a study group and a control group in the A-PRF group. The implants were placed symmetrically to the right and left of the midline by the same physician provided that they were in the same jaw.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group in which the patients were included was determined by pulling the closed envelope just before the surgery. Test side was determined by tossing a coin after the implant cavities were prepared but before the implants were placed. The examiners who carried out the measurements and analyzes were unaware of the study and the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A-PRF Test Group (Experimental): Advanced Platelet Rich Fibrin liquid applied into the implant cavity and implant surface. That is the only difference between A-PRF control group and A-PRF test group.
  Interventions: Procedure: Advanced platelet rich fibrin (A-PRF)
- CGF Test Group (Experimental): Concentrated growth factor liquid applied into the implant cavity and implant surface. That is the only difference between CGF control group and CGF test group.
  Interventions: Procedure: Concentrated growth factor(CGF)
- A-PRF Control Group (Experimental): Dental implant applications were made with traditional methods.
  Interventions: Procedure: Control side of advanced platelet rich fibrin study group
- CGF Control Group (Experimental): Dental implant applications were made with traditional methods.
  Interventions: Procedure: Control side of concentrated growth factor study group

INTERVENTIONS:
Procedure: Concentrated growth factor(CGF) — Concentrated growth factor(CGF) liquid applied to the implant cavity and implant surface.
  Arms: CGF Test Group
Procedure: Advanced platelet rich fibrin (A-PRF) — Advanced platelet rich fibrin (A-PRF) liquid applied to the implant cavity and implant surface.
  Arms: A-PRF Test Group
Procedure: Control side of concentrated growth factor study group — Traditional implant methods applied.
  Arms: CGF Control Group
Procedure: Control side of advanced platelet rich fibrin study group — Traditional implant methods applied.
  Arms: A-PRF Control Group

SUMMARY:
In this study, concentrated growth factor obtained by centrifuging the patient's own blood and advanced platelet-rich fibrin liquids were applied to the implant cavity and surface. Thus, it was aimed to ensure that the osseointegration process would start earlier by ensuring a faster arrival of growth factor and healing mediators in the region, and thus, the time waited for the osseointegration process and the loading of the superstructure would be shortened.

In this split-mouth study, a total of 32 patients including two separate study groups in different patients and a control group were included. While the CGF liquid was applied to the implant cavities and surfaces prepared in the study group of 16 patients, A-PRF liquid was applied to the study group of the other 16 patients. Conventional implant application was performed in the control groups of both groups. The torque values during the implantation were also recorded, and Resonance Frequency measurements were performed immediately after implantation with the Penguin RFA device and at postoperative weeks 2, 4, 6 and 12.

DETAILED DESCRIPTION:
This study was conducted in accordance with the Helsinki declaration on 32 patients who applied to Hatay Mustafa Kemal University Faculty of Dentistry Department of Oral and Maxillofacial Surgery to have dental implants in order to fix their missing teeth. 2 implants with appropriate sizes and diameters were applied to each patient according to the condition of the recipient bone in order to ensure standardization. It was aimed to ensure that the primary stabilization of the implant would not be affected locally by applying implants to the sites with similar bone density. The implants were placed symmetrically to the right and left of the midline by the same physician provided that they were in the same jaw.

Some conditions were required for the inclusion of patients in the study, which were:

* Having no systemic disorder,
* Not being pregnant or breastfeeding,
* Having no smoking habit,
* Lack of continuous drug use due to chronic disease,
* No infection in the implant site and adjacent teeth,
* No previous implant or any augmentation procedure in the implant site,
* Adequate bone height and thickness of the implant site,
* The patient's acceptance and signing the informed consent form specific to study describing the aim, duration, advantages and possible complications of the study.

Among the inclusion criteria in the study, no distinction was made between men and women, and the patients without these criteria were not included in the study.

This study evaluating the effects of advanced platelet-rich fibrin and concentrated growth factor liquids on dental implant osseointegration was planned as a randomized, clinical controlled and prospective study. A total of 32 patients included in this study were divided into two groups of 16. It was planned to apply 2 implants to each patient and to evaluate each patient as one side as the control and the other as the study group. In other words, while there was a study group and a control group in the CGF group, there was also a study group and a control group in the A-PRF group. In the first group, it was planned to wash the surface of one of the implants to be applied and the inside of the socket where the implant would be placed with the CGF liquid obtained by centrifuging the patient's own blood, and to apply a standard implant procedure without any application to the socket and surface of the other implant to be applied.

In the second group, the surface of the implant in the study group the inside of the socket where the implant would be placed were washed with the A-PRF liquid obtained by centrifuging the patient's own blood, and standard conventional implant procedure was applied without any application to the implant socket and surface in the control group.

Obtaining the CGF Liquid:

Sterile, single use, anticoagulant-free tube (Vacutest®, Arzergrande-Italy), syringe sets for taking blood, skin disinfectant, centrifuge device produced suitable for tubes (MEDIFUGE, Italy), and a special sterile container for obtaining the serum part of the concentrated growth factor were used for the preparation of the concentrated growth factor. 2 x 9 cc. venous blood samples taken intravenously from the patients were placed in the centrifuge machine in tubes without shaking.

By operating the centrifuge in CGF mode, the device accelerated with an acceleration of 30 seconds and was centrifuged for 2 minutes at 2700 rpm, 4 minutes at 2400 rpm, 4 minutes at 2700 rpm and 3 minutes at 3000 rpm, and then the device stopped with an acceleration of 36 seconds. The process and periods of change of all this turnover rate are automatically adjusted by the device. After the centrifugation process, 3 layers occur in the tube. These layers were platelet-poor plasma layer at the top, red blood cell layer at the bottom, and concentrated growth factor layer in the middle, respectively. The concentrated growth factor formed was separated from the red blood cell layer in the lower layer with the help of scissors by holding it with the help of a hemostat. However, during the separation process, the part containing CD34+ stem cells was kept below the concentrated growth factor. Then, the CGF was placed in a special sterile perforated container, pressed in the container and turned into a membrane. Thus, the serum part of CGF was obtained by means of the holes in the container.

Obtaining the A-PRF Liquid:

Sterile, single use, anticoagulant-free A-PRF tube, centrifuge device Duo centrifuge (Process for PRF, France) produced suitable for these tubes, and a special sterile container for obtaining the serum part of the A-PRF were used for the preparation of the A-PRF.

2x10 cc. venous blood samples taken intravenously from the patients were placed in the centrifuge device without shaking, and centrifugation was set at 1300 rpm for 14 minutes. While the A-PRF clot formed after the centrifugation was separated from the lower red blood cell layer with the help of a hemostat, attention was paid not to remove this layer completely. Then, this fibrin clot was pressed in a special sterile perforated contained and A-PRF liquid was obtained.

Surgical Procedure:

All surgical procedures were performed as a double-blind study by the same surgical team. After providing local anesthesia in the region, a crestal incision was made in the area to be implanted using a scalpel number 15, and then, full-thickness mucoperiosteal flap was removed. After the study and control groups were randomly determined, the implant socket was prepared in appropriate size and diameter according to the surgical kit of the implant system (Nucleoss T6, Turkey). In the study group of the concentrated growth factor, the surface of the implant and the socket where the implant would be placed were washed with the CGF liquid and placed in the implant socket without deterioration of sterility (Figure 2). The implant in the control group was placed in its socket with the standard implant procedure without any procedure. Similarly, the implants were placed in their sockets as stated above in the study and control groups of the advanced platelet-rich fibrin. After all the implants in the study and control groups were placed in the socket, the adjustable ratchet torque on the carrying piece on it placed in 1 mm subcrestal position with a wrench in the buccal and lingual/palatinal area. Thus, torque values were also recorded. The ratchet wrench measuring torque values in the range of 10-50 N specially produced by Nucleoss company was used for this study. After the implant application, a suitable healing cap was placed on all implants and the wound edges were sutured with mucoperiosteal flap 3-0 silk suture so that the healing caps would not be covered. The patients were recommended to apply a cold compress after the surgical procedure. After the operation, Amoxicillin + Clavulanic acid 1 g (Augmentin) one tablet twice a day for 7 days, Analgesic and anti-inflammatory Dexketoprofen 25 mg (Arveles) one tablet twice a day for 5 days, and 0.12% chlorhexidine mouthwash (Kloroben) 3 times a day were prescribed. The patients were informed about the points to be considered after the procedure.

Resonance Frequency Analysis Measurement:

Penguin Resonance Frequency Analysis (RFA) (Integration Diagnostics Sweden AB) device and MulTipeg, a transducer suitable for the implant the investigators would place, were used to obtain the Implant Stability Quotient (ISQ) values of the implants by resonance frequency analysis and to evaluate their stability. With the help of a MulTipeg carrier, it was tightened and placed on the implant until resistance was encountered (manual tightening torque of approximately 3-5 Ncm). During the use of Penguin, measurement is made without touching the tip of the probe to the MulTipeg, therefore, it does not require any contact. Furthermore, it is completely non-invasive and the patient does not feel anything during the measurement, which takes a few seconds. The stability is indicated on the implant by the ISQ value. RFA values were measured for a total of 5 times, namely immediately after implantation and at postoperative weeks 2, 4, 6 and 12. In order to obtain the ISQ value, the arithmetic mean of the numerical values obtained by measuring the mesio-distal and bucco-lingual total five times in two directions perpendicular to each other was recorded as ISQ unit.

ELIGIBILITY:
Inclusion Criteria:

* - Having no systemic disorder,
* Not being pregnant or breastfeeding,
* Having no smoking habit,
* Lack of continuous drug use due to chronic disease,
* No infection in the implant site and adjacent teeth,
* No previous implant or any augmentation procedure in the implant site,
* Adequate bone height and thickness of the implant site,
* The patient's acceptance and signing the informed consent form specific to our study describing the aim, duration, advantages and possible complications of the study.

Among the inclusion criteria in the study, no distinction was made between men and women, and the patients without these criteria were not included in the study.

Ages: 38 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Torque values | Immediately after surgery
  The torque values measured immediately after the implant placement.
Resonance Frequency Analysis-I | Immediately after surgery
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-II | Second week
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-III | Fourth week
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-IV | Sixth week
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.
Resonance Frequency Analysis-V | Twelfth week
  Resonance frequency analysis is a method used to determine the primer stability in dental implants.

CONTACTS AND LOCATIONS:
Locations (1):
- Ugur Can Unlugenc, Hatay, Mustafa Kemal University Hatay, Turkey, 31060, Turkey (Türkiye)